CLINICAL TRIAL: NCT02093962
Title: A Randomized Phase 2, Double-blind, Placebo-controlled, Multi-center Study Comparing Pemetrexed in Combination With TH-302 vs. Pemetrexed in Combination With Placebo as Second-line Chemotherapy for Advanced Non-Squamous, Non-Small Cell Lung Cancer
Brief Title: Study of TH-302 or Placebo in Combination With Pemetrexed in Patients With Non-squamous Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: At the interim analysis, the futility boundary was not met and the study was stopped due to insufficient efficacy.
Sponsor: ImmunoGenesis (Industry)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TH-CR-415
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: TH-302; TH-CR-415; Pemetrexed; Non-small cell lung cancer; Lung cancer; Evofosfamide
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TH-302 and pemetrexed (Experimental): TH-302 in combination with pemetrexed
  Interventions: Drug: TH-302 combination with pemetrexed
- Placebo and pemetrexed (Active Comparator): Matching placebo in combination with pemetrexed
  Interventions: Drug: Matched placebo in combination with pemetrexed

INTERVENTIONS:
Drug: TH-302 combination with pemetrexed — 400 mg/m2 of TH-302 will be administered by IV infusion over 30 - 60 minutes on Day 1 and Day 8 of a 21-day cycle.
  Pemetrexed (500 mg/m2) will be administered as an IV infusion on Day 1 two - four hours after TH-302 administration.
  Arms: TH-302 and pemetrexed
Drug: Matched placebo in combination with pemetrexed — Matched placebo will be administered by IV infusion over 30 - 60 minutes on Day 1 and Day 8 of a 21-day cycle.
  Pemetrexed (500 mg/m2) will be administered as an IV infusion on Day 1 two - four hours after placebo administration.
  Arms: Placebo and pemetrexed

SUMMARY:
The purpose of this study is to determine whether TH-302 in combination with pemetrexed is safe and effective in the treatment of non-squamous non-small cell lung cancer.

DETAILED DESCRIPTION:
TH-302 is designed to target the hypoxic regions of tumors which are generally located distant from tumor vessels. Pemetrexed has poor tissue penetration and targets the regions of tumors that are located in proximity to the tumor vessels. The presence of hypoxia in solid tumors is associated with a more malignant phenotype and resistance to chemotherapy. The hypoxia-activated prodrug, TH-302, is designed to selectively target the hypoxic microenvironment. There is evidence supporting the presence of hypoxia in NSCLC lesions based on a hypoxia PET study. Combining pemetrexed with TH-302 may enable the targeting of both the normoxic and hypoxic regions of NSCLC lesions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Histologically or cytologically confirmed stage IIIB or IV NSCLC with non-squamous histology
* Recurrent or progressive disease after one prior platinum-based non-pemetrexed chemotherapy treatment for advanced disease with or without maintenance
* Neoadjuvant/adjuvant cytotoxic chemotherapy initiated < 12 months prior to study randomization will be counted as one prior treatment
* Neoadjuvant/adjuvant cytotoxic chemotherapy initiated ≥ 12 months prior to study randomization will not be counted as one prior chemotherapy treatment
* Use of targeted agents (e.g., monoclonal antibodies or kinase inhibitors) will not be counted as a prior chemotherapy treatment
* Patients with known EGFR-activating mutations or ALK rearrangements should have received treatment with a targeted kinase inhibitor (e.g., erlotinib, crizotinib) and no longer be considered as a candidate for such treatment
* Measurable disease according to RECIST 1.1
* ECOG performance status 0-1
* Resolution to Grade ≤ 1 Adverse Events, of all clinically significant toxic effects of prior therapy
* Adequate hematologic, hepatic, cardiac, and renal function
* Female patients of childbearing potential must have a negative serum or urine pregnancy test, whichever is considered standard by the institution

Exclusion Criteria:

* Diagnosis of small cell carcinoma of the lung, squamous cell carcinoma of the lung or NSCLC NOS
* Prior therapy with pemetrexed
* Inability or unwillingness to take folic acid, vitamin B12 supplementation or corticosteroids
* Inability to discontinue non-steroidal anti-inflammatory drugs for 5 days (long half-life) or for 2 days (short half-life, if CrCL <80 mL/min) before pemetrexed dosing and until 2 days after pemetrexed dosing
* Leptomeningeal disease or any untreated or symptomatic brain metastases, unless the following criteria are met:

  * brain metastases are stable and have been previously treated with either whole-brain radiotherapy or gamma-knife surgery
  * steroids are currently not required and more than 14 days since last steroid treatment
* Symptomatic pleural effusion (> CTCAE Grade 1 dyspnea) that is not amenable to drainage
* Treatment with other systemic anticancer therapy within 4 weeks prior to the first dose of study medication
* Treatment with full field radiation therapy within 4 weeks or limited field radiation therapy within 2 weeks prior to the first dose of study medication
* Major surgery within 4 weeks or minor surgery within 2 weeks prior the first dose of study medication
* Elective or a planned major surgery while on study treatment
* Radiation therapy to greater than 25% of the bone marrow
* Clinically significant active infection (e.g. tuberculosis, viral hepatitis, HIV)
* Any other serious uncontrolled medical disorders or psychological conditions that may interfere with study conduct
* Concurrent active malignancy other than adequately treated basal cell or squamous cell carcinoma of the skin or pre-invasive carcinoma of the cervix.
* Pregnant or breast feeding
* Patients who are taking medications that prolong QT interval and have a risk of Torsades de Pointes (Appendix F) or who have a history of long QT syndrome
* Patients who are taking medications that are strong inducers or inhibitors of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2014-06; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tillman Pearce, MD, Study Chair — Threshold Pharmaceuticals; Jonathan Goldman, MD, Principal Investigator — UCLA-Dept of Medicine a Div of Hem/Onc
Locations (80):
- United States (29):
  - UAB Cancer Center, Birmingham, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - California Cancer Center, Encinitas, California
  - California Cancer Center Associates, Fresno, California
  - UCLA-Department of Medicine a Division of Hem/Onc, Los Angeles, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - VA Eastern Colorado Healthcare System, Denver, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Cancer Specialists of North Florida - CBO, Jacksonville Beach, Florida
  - AMPM Research, Miami, Florida
  - Research Medical Center, Kansas City, Kansas
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - St. Joseph Mercy Ann Arbor Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Clinical Research Alliance, New York, New York
  - Montefire-Einstein Center for Cancer Care, The Bronx, New York
  - Durham VA Medical Center, Durham, North Carolina
  - W.G. (Bill) Hefner VA Medical Center, Salisbury, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - DORN VA Medical Center, Columbia, South Carolina
  - Regional Cancer Care Institute at Regional Health, Rapid City, South Dakota
  - Associates in Oncology & Hematology, Chattanooga, Tennessee
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Oncology Consultants, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - Fpr Belvoir Community Hospital, Fort Belvoir, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
- Czechia (4):
  - Hospital Na Bulovce, Department of Pneumology and Thoracic Surgery, Libeň
  - General Univesity Hospital in Prague, Clinic of Oncology, Prague
  - Thomayer Hospital, Clinic of Pneumology, Prague
  - Regional Hospital T. Bta, Department of Pneumology, Zlín
- Germany (8):
  - Asklepios Fachkliniken Munchen-Gaunting, Gauting, Bavaria
  - Marien Hospital Herne, Herne, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin;, Berlin
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Lungen Clinic Grosshandsdorf GmbH, Großhansdorf
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Städtisches Klinikum München - Klinikum Bogenhausen, München
  - Universitätsklinikum Ulm; Zentrum für Innere Medizin, Ulm
- Greece (4):
  - IASO General, Oncology Unit, Athens
  - Attikon University General Hospital, Athens
  - Department of Medical Oncology, Heraklion
  - University General Hospital of Patras, Oncology Unit, Pátrai
- Hungary (6):
  - Koranyi National Institute of TBC and Pulmonology, 14th Dept of Pulmonology, Budapest
  - Koranyi National Institute of TBC and Pulmonology, 6th Department of Pulmonology, Budapest
  - Koranyi National Institute of TBC and Pulmonology, 8th Department of Pulmonology, Budapest
  - University of Debrecen, Medical and Health Science Center, Department of Pulmonology, Debrecen
  - Csongrad County Hospital of Chest Diseases, Deszk
  - Hetenyi Geza Hospital, Department of Oncology, Szolnok
- Italy (10):
  - "Mater Salutis" Hospital - Operative Unit of Oncology, Verona, Legnago
  - A.O.U.S. Luigi GonzagaUniversity Hospital, Orbassano, Torino
  - Hospital Bellaria "Carlo Alberto Pizzardi" - Operative Unit of Oncology, Bologna
  - IRCCS Azienda Ospedallera Universitaria San Martino-IST-Istituto Nazionale per la Ricerca sul Cancro, Genova
  - European Institute of Oncology (IEO) - Medical Care Unit, Milan
  - S. Gerardo Hospital - Complex Structure of Medical Oncology, Monza
  - Azienda Ospedaliera Universitaria Policlinico della Seconda Universita di Napoli, Napoli
  - University Hospital of Pisa, Department of Cardothoracic Surgery, Operative unit of Pneumology, Pisa
  - "Santa Maria degli Angeli" - Hospital - Complex Operative Unit of Oncology, Pordenone
  - San Camillo-Forlanini Hospital - U.O.C. Pneumologia Oncologica 1, Rome
- Poland (3):
  - Med-Polonia Sp. z o.o., Poznan
  - L. Rydygier Provencial Hospitals in Torun, Dept. of Tumors Chemotherapy, Torun
  - Maria Sklodowska-Curie Institute of Oncology in Warsaw, Warsaw
- Romania (3):
  - Oncology Centre "Sf. Nectarie", Craiova, Dolj
  - Pro. Dr. Alex Trestioreanu Institute of Oncology, Bucharest
  - Prof. Dr. Ioan Chiricuta Institute of Oncology, Cluj-Napoca
- Russia (7):
  - Republican Clinical Oncology Center under the Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Russian Oncology Research Center n.a. N.N. Blokhin under the Russian Academy of Medical Sciences, Moscow
  - Blokhin Russian Oncology Research Center, Moscow
  - State Healthcare Institution: Nizhny Novgorod Regional Oncology Center, Nizhny Novgorod
  - St. Petersburg Clinical Center for Applied Special Medical Services (Oncology), Saint Petersburg
  - St. Petersburg 1st State Medical University n.a.I.P. Pavlov under the Ministry of Healthcare of the Russian Federation, Saint Petersburg
  - City Clinical Oncology Center, Oncology Department (Thoracic Oncology), Saint Petersburg
- Spain (6):
  - General University Hospital Gregorio Maranon, Dept. of Oncology, Madrid
  - Jimenez Diaz Foundation, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - University Hospital Virgen de Valme, Seville
  - Dr. Peset University Hospital, Dept. of Oncology, Valencia
  - Hospital Universitario La Fe, Servicio de Oncologia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- TH-302 and Pemetrexed: TH-302 in combination with pemetrexed
  TH-302 combination with pemetrexed: 400 mg/m2 of TH-302 will be administered by IV infusion over 30 - 60 minutes on Day 1 and Day 8 of a 21-day cycle.
  Pemetrexed (500 mg/m2) will be administered as an IV infusion on Day 1 two - four hours after TH-302 administration.
- Placebo and Pemetrexed: Matching placebo in combination with pemetrexed
  Matched placebo in combination with pemetrexed: Matched placebo will be administered by IV infusion over 30 - 60 minutes on Day 1 and Day 8 of a 21-day cycle.
  Pemetrexed (500 mg/m2) will be administered as an IV infusion on Day 1 two - four hours after placebo administration.
Period: Overall Study
Arm/Group | TH-302 and Pemetrexed | Placebo and Pemetrexed
Started | 134 | 131
Received Treatment | 130 | 130
Completed | 0 | 0
Not Completed | 134 | 131

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TH-302 and Pemetrexed | Placebo and Pemetrexed | Total
Number analyzed (Participants) | 134 | 131 | 265
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 85 | 166
  >=65 years | 53 | 46 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 57 | 115
  Male | 76 | 74 | 150
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 3 | 6
  White | 130 | 126 | 256
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: To assess the efficacy of pemetrexed in combination with TH-302 as determined by overall survival in patients with advanced non-squamous NSCLC in the second-line chemotherapy setting compared with pemetrexed in combination with placebo
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | TH-302 and Pemetrexed | Placebo and Pemetrexed
Number analyzed (Participants) | 134 | 131
Participants | 51 | 49

ADVERSE EVENTS:
Arm/Group | TH-302 and Pemetrexed | Placebo and Pemetrexed
Serious Adverse Events (participants affected / at risk) | 52/130 | 72/130
Other Adverse Events (participants affected / at risk) | 130/130 | 130/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 and Pemetrexed (N=130) | Placebo and Pemetrexed (N=130)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 7 (11)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Quadriplegia (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 and Pemetrexed (N=130) | Placebo and Pemetrexed (N=130)
Anaemia (Blood and lymphatic system disorders) | 40 (56) | 50 (80)
Neutropenia (Blood and lymphatic system disorders) | 24 (70) | 30 (83)
Thrombocytopenia (Blood and lymphatic system disorders) | 10 (19) | 25 (47)
Decreased appetite (Metabolism and nutrition disorders) | 20 (27) | 17 (27)
Headache (Nervous system disorders) | 16 (20) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (23) | 19 (21)
Diarrhoea (Gastrointestinal disorders) | 16 (24) | 23 (43)
Nausea (Gastrointestinal disorders) | 37 (79) | 40 (76)
Stomatitis (Gastrointestinal disorders) | 18 (26) | 24 (45)
Vomiting (Gastrointestinal disorders) | 17 (20) | 25 (34)
Asthenia (General disorders) | 19 (30) | 28 (48)
Fatigue (General disorders) | 25 (33) | 33 (44)
Alanine aminotransferase increased (Investigations) | 16 (27) | 17 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No